CLINICAL TRIAL: NCT02833337
Title: Morphological Pattern of the Atrophic Posterior Maxillae
Status: Completed | Type: Observational
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Sponsor
Other Study IDs: 52/2012
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-08

CONDITIONS: Bone Deficiency, Posterior Maxillae
Keywords: Bone; Maxilla; Cone-Beam Computed Tomography; Regeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Radiation: Cone-beam computed topography — This study used a retrospective database of preexisting data that included patients treated as part of routine periodontal and oral surgery therapy for each patient's needs. All the patients signed an inform consent approving using their radiographic data for research purposes.

SUMMARY:
Overcoming the vertical and horizontal bone deficiency in the posterior maxillae are considered as the most challenging scenarios for implant-supported oral rehabilitation in modern implant dentistry. Therefore, a comprehensive and precise understanding of such anatomical structures are needed to avoid potential complications that ultimately might jeopardize the treatment outcome.

Cone-beam computerized tomography (CBCT) offers some advantages to conventional CT-scan such as lower-dose radiation with high isotropic spatial resolution and cost. Therefore, it offers a viable and reliable tool to study anatomical structures such as the posterior atrophic maxillae

ELIGIBILITY:
* Images were included if:

  1. Pristine maxillary posterior atrophic ridges (between premolars and molars) as a result of missing single or multiple teeth for over than 12 months.
  2. Residual ridge height (RH) was < 10 mm.
  3. Presence of teeth adjacent to or opposing the edentulous area so the location of the edentulous ridges corresponding to the tooth site could be identified.
  4. The maxillary sinus to be measured was visible from its floor to at least 15 mm from the alveolar crest of the edentulous ridge.
* Images were excluded if:

  1. Images were unclear or incomplete due to scattering or other reasons
  2. Edentulous ridge height was more than 10 mm
  3. Ridge preservation/augmentation simultaneous/delayed to tooth extractions
  4. Grafted maxillary sinus for implant-supported prosthesis
  5. The location of the edentulous ridge cannot be determined
  6. Implants or other prosthetic device restoring the posterior ridge
  7. Presence of sinus pathology that made the measurement impossible
  8. The outline of the edentulous ridge cannot be identified due to low 'grey scale' density

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study used a retrospective database of preexisting data that included patients treated as part of routine periodontal and oral surgery therapy for each patient's needs. All the patients signed an inform consent approving using their radiographic data for research purposes.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Florencio Monje Gil, Badajoz, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- Consecutive Individuals: Consecutive individuals explored via cone-beam computed tomography to evaluate the anatomical features
Period: Overall Study
Arm/Group | Consecutive Individuals
Started | 180
Completed (180 completed) | 180
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Consecutive Individuals
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 110
  >=65 years | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 100
Region of Enrollment [Number; unit: participants]
  Spain | 180

OUTCOME MEASURES:

1. Primary Outcome: Lateral Wall Thickness
Description: Thickness measured in mm of the lateral aspect of the maxillary sinus
Time Frame: One month
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Consecutive Individuals
Number analyzed (Participants) | 180
mm | 161 (11)

ADVERSE EVENTS:
Time Frame: No adverse events were monitored
Description: No adverse events were monitored given the nature of the study (i.e., cross-sectional radiographic analysis)
Groups:
- No Adverse Events Were Monitored: Adverse events were not monitored
Arm/Group | No Adverse Events Were Monitored
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes